CLINICAL TRIAL: NCT01461460
Title: A Phase 1 Blinded, Placebo-controlled Crossover Study to Evaluate the Effects of Oral TR 701 Free Acid on the Electrocardiogram
Brief Title: A Thorough QT Study of TR-701free Acid (FA) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1986-029; TR701-115 (Other: TriusRX unique ID)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteer
Keywords: volunteer
MeSH Terms: interventions — tedizolid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moxifloxacin 400 mg (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg
- TR-701 FA 1200 mg (Experimental)
  Interventions: Drug: TR-701 FA 1200 mg
- TR-701 FA 200 mg plus Placebo (Experimental)
  Interventions: Drug: TR-701 FA 200 mg plus Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TR-701 FA 1200 mg — 6 tablet of T-701 FA
  Other Names: Tedizolid
  Arms: TR-701 FA 1200 mg
Drug: Moxifloxacin 400 mg — 1 tablet 400 mg Moxifloxacin
  Arms: Moxifloxacin 400 mg
Drug: TR-701 FA 200 mg plus Placebo — 1 tablet of TR-701 FA with 5 tablet placebo
  Other Names: Tedizolid
  Arms: TR-701 FA 200 mg plus Placebo
Drug: Placebo — 6 placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of oral TR-701 free acid (FA) versus placebo on QTcF.

DETAILED DESCRIPTION:
To assess the effects of a single therapeutic (200 mg) and supratherapeutic of oral TR-701 free acid (FA) versus placebo on QT interval corrected for heart rate using Fridericia's formula (QTcF) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 45 years of age, inclusive.
* Healthy males and females with no clinically significant abnormalities.
* Body mass index ≥18.0 kg/m2 and ≤30.0 kg/m2

Exclusion Criteria:

* Sustained supine systolic blood pressure >140 or <100 mmHg or a diastolic blood pressure >90 or <60 mmHg at the Screening and Day 1 Visit.
* Abnormal ECG at Screening or Day -1 Visits indicating a second or third-degree atrioventricular block, or QRS >110 msec, QTcF >450 msec for males and >470 msec for females, PR interval >200 msec, or any rhythm other than sinus rhythm which is interpreted by the Investigator as clinically significant - History of unexplained infections or current signs of infection
* History of risk factors for Torsades de Pointes, including unexplained syncope, known Long QT Syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, hypomagnesemia, or family history of Long QT Syndrome or Brugada Syndrome

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2011-12-23 (Actual); Study Completion 2011-12-23 (Actual)

PRIMARY OUTCOMES:
QTcF Change from Baseline | 24 Hours
  Time-matched, placebo adjusted change from the baseline QTcF (ΔΔQTcF).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator, Dallas, Texas, United States

REFERENCES:
- [Background] Flanagan S, Litwin J, Fang E, Prokocimer P. Effects of therapeutic and supratherapeutic doses of oral tedizolid phosphate on cardiac repolarisation in healthy volunteers: a randomised controlled study. Int J Antimicrob Agents. 2016 Jul;48(1):33-40. doi: 10.1016/j.ijantimicag.2015.12.015. Epub 2016 Jun 2. PMID 27342387